CLINICAL TRIAL: NCT02032810
Title: A Phase 1 Study of HDAC Inhibitor Panobinostat (LBH 589) Administered in Combination With Ipilimumab in Subjects With Unresectable Stage III or Stage IV Melanoma
Brief Title: Phase I of Histone Deacetylase (HDAC) Inhibitor Panobinostat With Ipilimumab With Unresectable III/IV Melanoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MCC-17439
Record Dates: First submitted 2014-01-08; First posted 2014-01-10 (Estimated); Results first posted 2019-07-02 (Actual); Last update posted 2023-01-20 (Actual); Status verified 2023-01

CONDITIONS: Melanoma; Skin Cancer
Keywords: Stage III Melanoma; Stage IV Melanoma; HDAC Inhibitor
MeSH Terms: conditions — Melanoma; Skin Neoplasms | interventions — Panobinostat; Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dose Escalation (Experimental): Dose Escalation of Panobinostat + Ipilimumab. Participants will be assigned to receive a certain dose of panobinostat (5, 10, 15, or 20 mg) along with a dose of ipilimumab of 3 mg per kg (mg/kg) of body weight.
  Interventions: Drug: Panobinostat; Drug: Ipilimumab

INTERVENTIONS:
Drug: Panobinostat — Participants will be assigned to receive a certain dose of panobinostat (5, 10, 15, or 20 mg). The dose of panobinostat will depend on the time point the participant enters the study and the side effects of other participants already on the study.
  Other Names: LBH 589
Drug: Ipilimumab — Dose of ipilimumab of 3 mg per kg (mg/kg) of body weight.
  Other Names: BMS-734016

SUMMARY:
The purpose of this study is to find out if an investigational drug called panobinostat can be given safely with another drug called ipilimumab. Investigators want to learn more about the side effects of this combination of drugs using different doses of panobinostat and the same dose of ipilimumab.

ELIGIBILITY:
Inclusion Criteria:

* Men and women ≥ 18 years old
* Participants must be ipilimumab naïve with progressive unresectable Stage III or Stage IV melanoma who are either treatment naïve or may have been treated with up to 3 prior treatments for melanoma (e.g., chemotherapy, biologic or targeted therapy or IL-2).
* Histologic or cytologic confirmation of stage III or stage IV melanoma
* Measurable disease at baseline as assessed by CT and/or MRI
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1
* Screening laboratory values must meet the following criteria: white blood count (WBCs) ≥ 2000/μL; Neutrophils ≥ 1500/μL; Platelets ≥ 100 x 10^3/μL; Hemoglobin ≥ 9.0 g/dL; Creatinine Serum creatinine ≤ 1.5 x upper limit of normal (ULN) or creatinine clearance > 40 mL/minute (using Cockcroft/Gault formula); aspartic transaminase (AST) ≤ 3 x ULN; alanine transaminase (ALT) ≤ 3 x ULN; Total Bilirubin ≤ 1.5 x ULN (except those with Gilbert Syndrome who must have total bilirubin < 3.0 mg/dL)
* Men and women of childbearing potential (WOCBP) must be using an acceptable method of contraception to avoid pregnancy throughout the study and for at least 12 weeks after the last dose of investigational product in such a manner that the risk of pregnancy is minimized. Women must have a negative serum pregnancy test within 72 hours prior to the start of investigational product.

Exclusion Criteria:

* Known or suspected brain metastasis, or brain as the only site of disease, with the following exceptions: controlled brain metastasis (no radiographic progression at least 4 weeks following radiation and/or surgical treatment, off steroids for at least 4 weeks, and have no new or progressing neurological signs or symptoms); history of prior malignancy with the exception of carcinoma in situ of the cervix or other malignancy diagnosed > 2 years ago that has undergone potentially curative therapy with no evidence of disease for the last ≥ 2 years and that is deemed by the investigator to be at a low risk of recurrence
* Active autoimmune disease or a history of known or suspected autoimmune disease with the exception of subjects with isolated vitiligo, treated thyroiditis or resolved childhood asthma/atopy
* Known human immunodeficiency virus (HIV), active hepatitis A, or hepatitis B or C infection
* History of any hepatitis (e.g., alcohol or non-alcohol steatohepatitis (NASH), drug- related, autoimmune)
* Evidence of active infection that requires anti-bacterial, anti-viral, or anti-fungal therapy ≤ 7 days prior to initiation of study drug therapy
* History of acute diverticulitis, or current chronic diarrhea
* Active peptic ulcer disease even if asymptomatic
* History of adrenal insufficiency (including subjects using replacement therapy)
* Prior organ allograft or allogeneic bone marrow transplantation
* Uncontrolled or significant cardiovascular disease including, but not limited to, any of the following: Myocardial infarction within the past 6 months; Uncontrolled angina within the past 6 months; Any history of clinically significant ventricular arrhythmias (such as ventricular tachycardia, ventricular fibrillation or Torsades de pointes). Controlled atrial fibrillation by itself is not an exclusion criterion.; Baseline corrected QT interval (QTc) interval greater than 500 milliseconds
* Baseline toxicities from prior anti-cancer treatments > Grade 1
* Inability to be venipunctured and/or tolerate venous access
* Any major surgery within 4 weeks or a diagnostic procedure (e.g. incision, needle biopsy) within 1 day of study drug administration
* Any current or recent (within 3 months) gastrointestinal disease that could potentially impact the ability to swallow and/or absorb study drug (i.e., gastrointestinal surgery, malabsorption syndrome)
* Diabetes mellitus uncontrolled by medication
* Known drug or alcohol abuse
* Presence of underlying medical condition that in the opinion of the Investigator or Sponsor could adversely affect the ability of the subject to comply with or tolerate study procedures and/or study therapy, or confound the ability to interpret the tolerability of combined administration of panobinostat and ipilimumab in treated subjects
* History of allergy to components of ipilimumab or panobinostat, or known allergy to other antibody therapies.
* WOCBP who are unwilling or unable to use an acceptable method to minimize the risk of pregnancy for the entire study period and for at least 12 weeks after the last dose of investigational product
* Women who are pregnant or breastfeeding
* Women with a positive pregnancy test on enrollment or prior to investigational product administration
* Sexually active fertile men not using effective birth control if their partners are WOCBP
* Exposure to any investigational drug within 4 weeks of study drug administration.
* Any anti-cancer therapy (e.g., chemotherapy, biologics, radiotherapy, or hormonal treatment) within 4 weeks or at least 5 half-lives (whichever is longer) of study drug administration
* Prior therapy with an anti-CTLA4 antibody or an HDAC inhibitor
* Concurrent chemotherapy, hormonal therapy, immunotherapy regimens, or radiation therapy, standard or investigational
* Prisoners or subjects who are involuntarily incarcerated
* Subjects who are compulsorily detained for treatment of either a psychiatric or physical (e.g., infectious disease) illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2014-01-07 (Actual); Primary Completion 2017-09-06 (Actual); Study Completion 2019-09-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nikhil Khushalani, M.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at Moffitt Cancer Center, November 2014 through November 2016.
Groups:
- Panobinostat 5 mg: Participants who received 5 mg of Panobinostat along with 3 mg Ipilimumab
- Panobinostat 10 mg: Participants who received Panobinostat 10 mg along with 3 mg Ipilimumab
Period: Overall Study
Arm/Group | Panobinostat 5 mg | Panobinostat 10 mg
Started | 6 | 11
Completed | 6 | 11
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Panobinostat 5 mg: Participants who received 5 mg of Panobinostat along with 3 mg Ipililumab
- Panobinostat 10 mg: Participants who received 10 mg of Panobinostat along with 3 mg Ipililumab
- Total: Total of all reporting groups
Arm/Group | Panobinostat 5 mg | Panobinostat 10 mg | Total
Number analyzed (Participants) | 6 | 11 | 17
Age, Continuous [Median (Full Range); unit: years] | 64 [56 to 75] | 66 [48 to 80] | 66 [48 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 4 | 9 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 6 | 10 | 16
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 6 | 11 | 17
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 6 | 11 | 17

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD)
Description: MTD and recommended Phase 2 dose (RP2D) of panobinostat (PAN), administered in combination with ipilimumab (IPI) in participants with unresectable Stage III or Stage IV melanoma.
  The goal is to enroll up to 36 patients for determination of the MTD, but will be successfully concluded earlier if 12 patients are accrued at the dose determined to be the MTD, with 3 dose limiting toxicities (DLTs).
  All participants who receive study any drug therapy will be evaluated for safety. Safety assessments will be based on medical review of adverse event reports and the results of vital sign measurements, physical examinations, and clinical laboratory tests. Triplicate 12-lead electrocardiograms (ECGs) will be collected prior to dosing on Day 1 of induction cycle 1. MTD of PAN in milligrams (mg), with IPI at 3 mg/kg.
Time Frame: Up to 36 months
Population: All participants
Measure: Number; unit: mg
Groups:
- Dose Escalation of Panobinostat, Plus Ipilimumab: Eligible participants with unresectable stage 3/4 MEL, up to 3 prior lines of therapy, and adequate laboratory values were treated with oral PAN 5 mg thrice weekly (TIW) plus IPI at 3 mg/kg IV every 3 weeks X 4 doses, followed by maintenance PAN until progression or intolerance. Using a modified Ji design, PAN dose escalation by 5 mg was planned in 3-12 participant cohorts up to a maximum dose of 20 mg TIW, without intra-participant dose escalation. Dose limiting toxicity (DLT) was assessed up to day 84 from start of therapy.
Arm/Group | Dose Escalation of Panobinostat, Plus Ipilimumab
Number analyzed (Participants) | 17
mg | 5

2. Secondary Outcome: Immune Related Overall Response Rate (ORR)
Description: Tumor response by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 and immune-related Response Criteria (irRC). RECIST: Best overall response from start of treatment until disease progression/recurrence. Immune-related Complete Response (irCR): Complete disappearance of all tumor lesions for at least 4 weeks from date of documentation of irCR. Immune-related Partial Response (irPR): Sum of the products of the 2 largest perpendicular diameters of all index lesions, measured and captured as the Sum of Product of Diameters (SPD) baseline. Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for Progressive Disease (PD), taking as reference the smallest sum longest diameter (LD) since the treatment started. Immune-related Progressive Disease (irPD): At least a 25% increase in the SPD of all index lesions and new measurable lesions (irSPD) over the nadir SPD calculated for the index lesions.
Time Frame: Up to 36 months
Measure: Count of Participants; unit: Participants
Arm/Group | Panobinostat 5 mg | Panobinostat 10 mg
Number analyzed (Participants) | 6 | 11
Participants
  Partial Response | 1 | 1
  Complete Response | 0 | 0
  Stable Disease | 3 | 3

3. Secondary Outcome: Progression Free Survival (PFS)
Description: Progression Free Survival (PFS): is defined for each participant as the time from first dosing to the first observation of disease progression or death due to any cause. If a subject has not progressed or died at the time of analysis, PFS will be censored on the date of the last disease assessment. PFS will be calculated by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1. Progressive Disease (PD) = 20% increase in the sum of the longest diameter of target lesions.
Time Frame: Up to 6 months
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Panobinostat 10 mg: Participants who received 10 mg of Panobinostat along with 3 mg of Ipilimumab
Arm/Group | Panobinostat 5 mg | Panobinostat 10 mg
Number analyzed (Participants) | 6 | 11
Months | 4.19 [1.68 to NA] — The high end of the range was not reached at time of analysis. | 1.81 [1.45 to NA] — The high end of the range was not reached at time of analysis.

4. Secondary Outcome: Overall Survival (OS)
Description: Overall survival: The time from randomization until death from any cause.
Time Frame: 36 months
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Panobinostat 5 mg: Participants who received 5 mg of Panobinostat along with 3 mg of Ipilimumab
- Panobinostat 10 mg: Participants who received 10 mg Panobinostat along with 3 mg Ipilimumab
Arm/Group | Panobinostat 5 mg | Panobinostat 10 mg
Number analyzed (Participants) | 6 | 11
Months | 25.91 [16.17 to NA] — The high end of the range was not reached at time of analysis. | 12 [6.58 to NA] — The high end of the range was not reached at time of analysis.

ADVERSE EVENTS:
Time Frame: 3 years, 9 months
Arm/Group | Panobinostat 5 mg | Panobinostat 10 mg
All-Cause Mortality (participants affected / at risk) | 1/6 | 0/11
Serious Adverse Events (participants affected / at risk) | 4/6 | 7/11
Other Adverse Events (participants affected / at risk) | 6/6 | 11/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Panobinostat 5 mg (N=6) | Panobinostat 10 mg (N=11)
Investigations - Other, Hypophysitis (Investigations) | 2 (2) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 1 (1)
Serum amylase increased (Investigations) | 0 (0) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Neoplasms - Other, basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Confusion (Psychiatric disorders) | 0 (0) | 2 (2)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 3 (3)
Renal and urinary disorders - Other, Hydronephrosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Rash maculopapular (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Hypotension (Vascular disorders) | 0 (0) | 2 (2)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Endocrine disorders - Other, Hypophysitis (Endocrine disorders) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 3 (3)
Nausea (Gastrointestinal disorders) | 1 (1) | 3 (4)
Vomiting (Gastrointestinal disorders) | 1 (1) | 2 (2)
Death NOS (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 3 (3)
Fever (General disorders) | 0 (0) | 2 (3)
Pain - Left groin/leg (General disorders) | 0 (0) | 1 (1)
Infections and infestations - Other, Tested positive for adenovirus (Infections and infestations) | 0 (0) | 1 (1)
Lung infection - Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Panobinostat 5 mg (N=6) | Panobinostat 10 mg (N=11)
Diarrhea (Gastrointestinal disorders) | 5 (6) | 9 (33)
Nausea (Gastrointestinal disorders) | 5 (8) | 8 (14)
Vomiting (Gastrointestinal disorders) | 4 (6) | 5 (12)
Abdominal pain (Gastrointestinal disorders) | 4 (4) | 3 (6)
Constipation (Gastrointestinal disorders) | 2 (2) | 4 (4)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 3 (4)
Bloating (Gastrointestinal disorders) | 1 (1) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 1 (1) | 1 (2)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 5 (11) | 10 (20)
Pain (General disorders) | 1 (1) | 3 (4)
Fever (General disorders) | 1 (1) | 2 (4)
General disorders and administration site conditions - Other (General disorders) | 2 (2) | 0 (0)
Malaise (General disorders) | 1 (1) | 1 (2)
Chills (General disorders) | 0 (0) | 1 (1)
Edema limbs (General disorders) | 0 (0) | 1 (1)
Flu like symptoms (General disorders) | 0 (0) | 1 (1)
Infusion related reaction (General disorders) | 1 (1) | 0 (0)
Localized edema (General disorders) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 3 (4) | 9 (10)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 3 (3)
Hyponatremia (Metabolism and nutrition disorders) | 1 (4) | 3 (9)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 0 (0) | 3 (8)
Lipase increased (Investigations) | 1 (4) | 2 (4)
Serum amylase increased (Investigations) | 1 (1) | 2 (2)
Weight loss (Investigations) | 0 (0) | 3 (3)
Creatinine increased (Investigations) | 2 (2) | 0 (0)
Investigations - Other (Investigations) | 2 (3) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Electrocardiogram QT corrected interval prolonged (Investigations) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Hematuria (Renal and urinary disorders) | 0 (0) | 3 (3)
Urinary frequency (Renal and urinary disorders) | 1 (1) | 2 (2)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 5 (6)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 2 (2) | 4 (5)
Endocrine disorders - Other (Endocrine disorders) | 2 (3) | 3 (6)
Adrenal insufficiency (Endocrine disorders) | 1 (1) | 0 (0)
Rash maculopapular (Skin and subcutaneous tissue disorders) | 1 (1) | 4 (5)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (3)
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (5) | 2 (4)
Dysgeusia (Nervous system disorders) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 1 (2) | 1 (3)
Amnesia (Nervous system disorders) | 1 (1) | 0 (0)
Concentration impairment (Nervous system disorders) | 1 (1) | 0 (0)
Nervous system disorders - Other (Nervous system disorders) | 0 (0) | 1 (2)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Confusion (Psychiatric disorders) | 1 (1) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 2 (2)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Cardiac disorders - Other (Cardiac disorders) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 0 (0) | 1 (3)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Conjunctivitis (Eye disorders) | 0 (0) | 1 (1)
Dry eye (Eye disorders) | 0 (0) | 1 (1)
Eye disorders - Other (Eye disorders) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 0 (0) | 1 (2)
Upper respiratory infection (Infections and infestations) | 0 (0) | 1 (2)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 2 (4)
Hot flashes (Vascular disorders) | 1 (1) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Postoperative hemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Immune system disorders - Other (Immune system disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-12-21): https://cdn.clinicaltrials.gov/large-docs/10/NCT02032810/Prot_SAP_000.pdf